CLINICAL TRIAL: NCT03048318
Title: Antegrade Arterial and Portal Flushing Versus Portal Flushing Only of the Liver Graft in Living Donor Liver Transplantation and Its Effects on Biliary Complications and Graft Function: A Randomized Control Study
Brief Title: Antegrade Arterial and Portal Flushing Versus Portal Flushing Only in LDLT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ILBS-ArterialFlush-001
Record Dates: First submitted 2017-01-31; First posted 2017-02-09 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-01

CONDITIONS: Biliary Complications; Graft Function, Delayed
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Intervention Model Description: Subsequent patients undergoing living donor liver transplant with right lobe grafts will be randomised
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arterial and Portal Flushing of Graft (Experimental): Back table flush of portal vein and graft artery
  Interventions: Procedure: Arterial Flushing; Procedure: Portal Flushing
- Portal Flushing only of Graft (Active Comparator): Back table flush of portal vein only
  Interventions: Procedure: Portal Flushing

INTERVENTIONS:
Procedure: Arterial Flushing
  Arms: Arterial and Portal Flushing of Graft
Procedure: Portal Flushing

SUMMARY:
Arterial flushing is a standard recommendation in deceased donor liver transplantation but not in living donor liver transplantation due to the risk of arterial intimal injury and short cold ischaemia time. There is recent evidence on benefit of retrograde arterial perfusion using hepatic venous occlusion and its benefits on post transplant cholestasis. However there is no data on antegrade arterial flushing.

DETAILED DESCRIPTION:
Biliary reconstruction has been labeled the "Achilles heel" of liver transplantation and is a common cause of postoperative morbidity and also mortality .Living donor liver transplantation (LDLT) has a higher incidence of biliary complications of up to 30% which is higher than Deceased Donor Liver Transplantation and does not seem to improve significantly with experience.The virtually unchanged incidence of biliary strictures suggests that they are not simply "technical" in origin, but probably represent a mucosa ischemic injury inherent in the transplantation procedure. The blood supply of the bile duct is mainly from the arterial system and skeletonisation of the duct during dissection impairs the blood supply rendering it ischemic.

Various donor maneuvers for better flushing and preserving peribiliary vascular plexus and biliary mucosa have been studied to decrease biliary complications. LDLT have advantages of haemodynamic stable donor and short cold ischemia but also has disadvantages of small graft size, small ducts, complicated reconstruction and absence of arterial flush. Conventional portal flush in animal livers could not remove warm blood from the arterial system and grafts without retrograde arterial flush had higher post operative bilirubin.With further studies in Living Donor Liver Transplant, it was concluded that retrograde flushing may ameliorate post operative cholestasis. There has not been data published on antegrade arterial flushing and its effect on biliary complications in Living Donor Liver Transplant. This study aims to compare back table graft arterial and portal flushing with portal flushing alone and evaluate biliary and arterial complications.

Arterial flushing has been made part of standard protocol at our institute and its safety established. There are centers which routinely perform back table arterial flush.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing living donor liver transplant for decompensated chronic liver disease with right lobe grafts only

Exclusion Criteria:

* Donor artery size less than 2 mm
* More than one donor artery
* GRWR <0.8
* ABO incompatible grafts
* Refusal to participate in the study
* Emergency transplants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Effects on biliary complications | Three months
  Occurence of biliary complication

SECONDARY OUTCOMES:
Hospital stay | 1 month
  Occurrence of complications
Morbidity | 1 month
Effect on graft function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rommel Sandhyav, MS, Principal Investigator — Institute of Liver and Biliary Sciences; Viniyendra Pamecha, MS, FRSS, FEBS, Principal Investigator — Professor; Senthil Kumar, MS, FRCS, Principal Investigator — Additional Professor; Shridhar Sasturkar, MS, MCh, Principal Investigator — Assistant Professor; Piyush Kumar Sinha, MS, MCh, Principal Investigator — Assistant Professor

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Pamecha V, Sandhyav R, Sinha PK, Bharathy KGS, Sasturkar S. Antegrade Arterial and Portal Flushing Versus Portal Flushing Only for Right Lobe Live Donor Liver Transplantation-A Randomized Control Trial. Transplantation. 2018 Apr;102(4):e155-e162. doi: 10.1097/TP.0000000000002088. PMID 29334530